CLINICAL TRIAL: NCT00843947
Title: Reduced Intensity Stem Cell Transplantation (RIST) for Patients With Hematological Malignancies Conditioned With Fludarabine and Busulfan
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200715041; UCD196
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Reduced Intensity Stem Cell Transplantation — Reduced Intensity Stem Cell Transplantation

SUMMARY:
This is a Phase II trial designed to evaluate the efficacy and toxicity of RIST, conditioned with fludarabine and busulfan, using G-CSF mobilized PBSC from an HLA-matched sibling or an unrelated volunteer donor. The primary endpoint of this study is day 100 TRM (Treatment Related Mortality). Secondary endpoints include response, engraftment times, acute and chronic GVHD, chimerism, toxicities, progression-free survival and overall survival.

Objectives

* To assess the efficacy and toxicity of Reduced Intensity Transplant (RIST) for patients with hematological malignancies, conditioned with fludarabine (Fludara®) and busulfan intravenous (Busulfex™).
* To evaluate progression-free survival and overall survival.
* To determine donor chimerism.
* To assess the risk of acute and chronic graft versus host disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed with (any of the following)

Disease Subtype Disease Status Leukemia Acute myelogenous leukemia (AML) Recurrent disease in remission* OR CR1 with poor-risk cytogenetics, antecedent hematological disease (i.e. myelodysplasia) or treatment-related leukemia Acute lymphoblastic leukemia (ALL) Recurrent disease in remission* OR CR1 with Philadelphia chromosome or poor risk cytogenetics Chronic myelogenous leukemia (CML) First or second chronic phase. There must be documented disease progression after imatinib mesylate (Gleevec) therapy OR documented lack of cytogenetic response 6 months post-imatinib initiation OR imatinib intolerance.

Patient - Inclusion criteria (Continued) Chronic lymphocytic leukemia (CLL) Recurrent disease after fludarabine-based therapy. Patients must have chemosensitive** disease at the time of relapse.

Lymphoma Recurrent Hodgkin's Lymphoma

Recurrent Non-Hodgkin's lymphoma (NHL) (Low, intermediate or high grade)

Transformed NHL Patients must have had prior autologous transplantation and received cytoreductive therapy at the time of relapse to achieve complete remission (CR) or CR/unconfirmed (CRu) as defined by the International Workshop

OR

Patient with relapsed disease and required >2 salvage regimens to achieve CR or CRu.

Multiple Myeloma Recurrent Myeloma Patients must have had prior autologous transplantation and demonstrate chemosensitivity** at the time of relapse Myelodysplastic Syndrome # RA/RARS RCMD/RCMD-RS RAEB-1 Patients must be transfusion-dependent and have International prostate symptom score (IPSS) of 1.5 or higher Advanced myeloproliferative disease Myelofibrosis with myeloid metaplasia; primary or evolved from other MPD Patient must be transfusion dependent or have evidence of progressive organomegaly or evidence of myelodysplasia

* remission is defined as morphological remission with bone marrow aspirate/biopsy showing <= 5% blasts within 4 weeks before the start of therapy. (Cytogenetic or molecular remission is not required)

  * In CLL, chemosensitivity is defined as greater than 50% reduction of wbc and lymphadenopathy. In MM, it is defined as greater than 50% reduction of M-component or plasma-cell marrow infiltration.

    * based on WHO classification system. Patients with RAEB-2 or del(5q) are excluded

      * 5-6/6 HLA-matched sibling or 9-10/10 matched unrelated donor
      * Age > 50 OR age 18-50, but have preexisting medical conditions, or have received prior therapy (i.e. prior) autologous transplantation) and are considered to be a too high a risk for conventional myeloablative transplantation

Exclusion Criteria:

* • Karnofsky performance status of less than 50%

  * Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy
  * Corrected pulmonary-diffusing capacity of less than 35%
  * A cardiac ejection fraction of less than 30%
  * A serologic evidence of infection with the human immunodeficiency virus
  * Inability to give informed consent
  * Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible
  * Decompensated liver disease with serum bilirubin > 2.0 mg/dl
  * Serum creatinine > 2.0 mg/dl
  * Uncontrolled active infection
  * Uncontrolled CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy and toxicity of Reduced Intensity Transplant (RIST) for patients with hematological malignancies, conditioned with fludarabine (Fludara®) and busulfan intravenous (Busulfex™) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of CA, Davis Cancer Center, Sacramento, California, United States